CLINICAL TRIAL: NCT03706040
Title: A Phase 2, Multicenter, Randomized, Placebo-Controlled, Double-Blind Study to Evaluate Risankizumab in Adult and Adolescent Subjects With Moderate to Severe Atopic Dermatitis
Brief Title: A Study to Evaluate Risankizumab in Adults and Adolescents With Moderate to Severe Atopic Dermatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M16-813; 2021-002203-34 (EudraCT Number)
Record Dates: First submitted 2018-10-11; First posted 2018-10-15 (Actual); Results first posted 2021-11-18 (Actual); Last update posted 2021-11-18 (Actual); Status verified 2021-10

CONDITIONS: Dermatitis
Keywords: Atopic dermatitis, Atopic dermatitis (atopic eczema)
MeSH Terms: conditions — Dermatitis; Dermatitis, Atopic | interventions — risankizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Placebo (Placebo Comparator): Participants randomized to receive placebo for 16 weeks in Period A followed by either risankizumab 150 mg or risankizumab 300 mg for 36 weeks in Period B.
  Interventions: Biological: Placebo; Biological: Risankizumab
- Risankizumab 150 mg (Experimental): Participants randomized to receive risankizumab 150 mg for 16 weeks in Period A followed by risankizumab 150 mg for 36 weeks in Period B.
  Interventions: Biological: Risankizumab
- Risankizumab 300 mg (Experimental): Participants randomized to receive risankizumab 300 mg for 16 weeks in Period A followed by risankizumab 300 mg for 36 weeks in Period B.
  Interventions: Biological: Risankizumab

INTERVENTIONS:
Biological: Placebo — subcutaneous (SC) injection
  Arms: Placebo
Biological: Risankizumab — subcutaneous (SC) injection
  Other Names: ABBV-066; BI 655066

SUMMARY:
The purpose of this study is to assess the safety and efficacy of risankizumab for the treatment of moderate to severe atopic dermatitis (AD) in adults and adolescents.

DETAILED DESCRIPTION:
This study includes a screening period of up to 35 days, a 16-week double-blind treatment period (Period A), and a 36-week double-blind treatment period (Period B).

Participants who meet eligibility criteria will be randomized at Baseline in a 2:2:1 ratio to one of 3 treatment groups: (1) risankizumab 150 mg, (2) risankizumab 300 mg, or (3) matching placebo. Randomization will be stratified by Baseline disease severity (Validated Investigator Global Assessment scale for Atopic Dermatitis [vIGA-AD] score of moderate [3] versus severe [4]) and geographic region (Japan versus rest of world).

At Week 16, participants in the placebo group will be re-randomized in a 1:1 ratio to receive either risankizumab 150 mg or 300 mg for the remainder of the study. Participants originally randomized to the risankizumab 150 mg or 300 mg arms will stay on their previously-assigned treatment through the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* adults who are ≥ 18 years old and, where locally permissible and approved, adolescent subjects who are at least 12 years old
* a diagnosis of atopic dermatitis (AD) with onset of symptoms at least 2 years prior to Baseline and subject meets Hanifin and Rajka criteria
* moderate to severe AD at the Baseline Visit
* history of inadequate response to previous topical corticosteroid and/or topical calcineurin inhibitor treatments or a medical inability to receive these treatments

Exclusion Criteria:

* prior exposure to any biologic immunomodulatory agent or Janus kinase (JAK) inhibitor
* concurrent treatment with systemic therapy for AD (biologic or non-biologic) or topical and/or phototherapy treatments

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2018-12-27 (Actual); Primary Completion 2020-10-28 (Actual); Study Completion 2021-04-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (65):
- United States (39):
  - UAB Department of Dermatology /ID# 211561, Birmingham, Alabama
  - Cognitive Clinical Trials /ID# 208895, Scottsdale, Arizona
  - Cosmetic Dermatology of Orange County /ID# 205801, Anaheim, California
  - Center for Dermatology Clinical Research /ID# 204950, Fremont, California
  - Integrative Skin Science and Research /ID# 212486, Sacramento, California
  - Cosmetic Laser Dermatology /ID# 210560, San Diego, California
  - Therapeutics Clinical Research /ID# 203422, San Diego, California
  - Colorado Center for Dermatology, PLLC /ID# 216260, Centennial, Colorado
  - Park Avenue Dermatology, PA /ID# 203378, Orange Park, Florida
  - MetroDerm ACC Research /ID# 205958, Atlanta, Georgia
  - Skin Care Physicians of Georgia /ID# 213188, Macon, Georgia
  - University Dermatology and Vein Clinic, LLC /ID# 210702, Darien, Illinois
  - The Indiana Clinical Trials Center /ID# 211618, Plainfield, Indiana
  - Tulane University /ID# 203214, New Orleans, Louisiana
  - DermAssociates /ID# 206189, Rockville, Maryland
  - Oakland Hills Dermatology /ID# 217453, Auburn Hills, Michigan
  - Duplicate_Great Lakes Research, Inc. /ID# 206447, Bay City, Michigan
  - Grekin Skin Institute /ID# 210485, Warren, Michigan
  - Skin Cancer and Dermatology Institute (SCDI) /ID# 213041, Reno, Nevada
  - Psoriasis Treatment Center of Central New Jersey /ID# 203203, East Windsor, New Jersey
  - Darst Dermatology /ID# 215100, Charlotte, North Carolina
  - Dermatologists of Southwest Ohio, Inc /ID# 215104, Mason, Ohio
  - Unity Clinical Research /ID# 217461, Oklahoma City, Oklahoma
  - Oregon Derm & Res. Ctr /ID# 202880, Portland, Oregon
  - Dermatologic SurgiCenter /ID# 208972, Drexel Hill, Pennsylvania
  - Dermdox Dermatology Centers, PC /ID# 212259, Hazleton, Pennsylvania
  - University of Pittsburgh MC /ID# 203296, Pittsburgh, Pennsylvania
  - Derm Assoc of Plymouth Meeting /ID# 208925, Plymouth Meeting, Pennsylvania
  - RI SkinDoc /ID# 203417, Johnston, Rhode Island
  - Omega Medical Research /ID# 216022, Warwick, Rhode Island
  - Health Concepts /ID# 203205, Rapid City, South Dakota
  - Rivergate Dermatology & Skin Care Center /ID# 203372, Goodlettsville, Tennessee
  - Arlington Research Center, Inc /ID# 215899, Arlington, Texas
  - Tekton Research, Inc. /ID# 211558, Austin, Texas
  - Center for Clinical Studies - Houston (Binz) /ID# 203383, Houston, Texas
  - Acclaim Dermatology /ID# 213026, Sugar Land, Texas
  - Virginia Dermatology & Skin Cancer Center /ID# 210154, Norfolk, Virginia
  - Dominion Medical Associates /ID# 212986, Richmond, Virginia
  - The Vancouver Clinic, INC. PS /ID# 202930, Vancouver, Washington
- Australia (6):
  - Woden Dermatology /ID# 204778, Phillip, Australian Capital Territory
  - St George Hospital /ID# 204780, Kogarah, New South Wales
  - Veracity Clinical Research /ID# 204786, Woolloongabba, Queensland
  - North Eastern Health Specialists /ID# 204785, Hectorville, South Australia
  - Skin Health Institute Inc /ID# 204779, Carlton, Victoria
  - Fremantle Dermatology /ID# 204784, Fremantle, Western Australia
- Canada (7):
  - Kirk Barber Research, CA /ID# 201046, Calgary, Alberta
  - Beacon Dermatology Inc /ID# 213003, Calgary, Alberta
  - University of Alberta Hospital - Division of Hematology /ID# 213008, Edmonton, Alberta
  - Medicor Research Inc /ID# 211274, Greater Sudbury, Ontario
  - Dr. Wei Jing Loo Medicine Prof /ID# 208849, London, Ontario
  - Lynderm Research Inc. /ID# 201050, Markham, Ontario
  - Dre Angelique Gagne-Henley M.D. inc. /ID# 208189, Saint-Jérôme, Quebec
- Japan (10):
  - Japan Organization of Occupational Health and Safety Chubu Rosai Hospital /ID# 213667, Nagoya, Aichi-ken
  - Kurume University Hospital /ID# 203139, Kurume-shi, Fukuoka
  - Nippon Medical School Musashi Kosugi Hospital /ID# 213961, Kawasaki-shi, Kanagawa
  - Nagaoka Red Cross Hospital /ID# 214140, Nagaoka-shi, Niigata
  - University of the Ryukyus Hospital /ID# 203974, Nakagami-gun, Okinawa
  - Osaka City University Hospital /ID# 203410, Osaka, Osaka
  - Hamamatsu University Hospital /ID# 203270, Hamamatsu, Shizuoka
  - Teikyo University Hospital /ID# 202884, Itabashi-ku, Tokyo
  - Tokyo Medical University Hospital /ID# 203647, Shinjuku-ku, Tokyo
  - Tokyo Medical University Hospital /ID# 204101, Shinjuku-ku, Tokyo
- Puerto Rico (3):
  - Dr. Samuel Sanchez PSC /ID# 213117, Caguas
  - Cruz-Santana, Carolina, PR /ID# 213229, Carolina
  - Clinical Research Puerto Rico /ID# 213118, San Juan

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols and clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing, please refer to the link below.
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous, independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Use Agreement (DUA). For more information on the process, or to submit a request, visit the following link.
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- [Derived] Tyring SK, Rich P, Tada Y, Beeck S, Messina I, Liu J, Huang X, Shumack S. Risankizumab in Patients with Moderate-to-Severe Atopic Dermatitis: A Phase 2, Randomized, Double-Blind, Placebo-Controlled Study. Dermatol Ther (Heidelb). 2023 Feb;13(2):595-608. doi: 10.1007/s13555-022-00876-x. Epub 2023 Jan 2. PMID 36588137

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adults and adolescents with moderate to severe atopic dermatitis (AD) with onset of symptoms at least 2 years before the Baseline visit were enrolled at 50 sites in the United States, Canada, Japan, and Australia.
  The study included a 16-week double-blind treatment period (Period A) followed by a 36-week double-blind treatment period (Period B).
Pre-assignment Details: Participants were randomized in a 2:2:1 ratio to risankizumab 150 mg, 300 mg, or placebo. Randomization was stratified by disease severity (Validated Investigator Global Assessment Scale for AD [vIGA-AD] moderate vs severe) and geographic region.
  At Week 16 participants in the placebo group were re-randomized in a 1:1 ratio to receive either risankizumab 150 mg or 300 mg in Period B. Participants originally randomized to risankizumab remained on their previously assigned treatment.
Groups:
- Period A: Placebo: Participants randomized to receive placebo by subcutaneous (SC) injection at Weeks 0 and 4 in Period A.
- Period A: Risankizumab 150 mg: Participants randomized to receive 150 mg risankizumab SC at Weeks 0 and 4 in Period A.
- Period A: Risankizumab 300 mg: Participants randomized to receive 300 mg risankizumab SC at Weeks 0 and 4 in Period A.
- Period B: Placebo / Risankizumab 150 mg: Participants initially randomized to placebo were re-randomized at Week 16 to receive 150 mg risankizumab SC at Week 16, Week 28, and Week 40 in Period B.
- Period B: Placebo / Risankizumab 300 mg: Participants initially randomized to placebo were re-randomized at Week 16 to receive 300 mg risankizumab SC at Week 16, Week 28, and Week 40 in Period B.
- Period B: Risankizumab 150 mg / Risankizumab 150 mg: Participants initially randomized to 150 mg risankizumab continued to receive 150 mg risankizumab SC at Week 16, Week 28, and Week 40 in Period B.
- Period B: Risankizumab 300 mg / Risankizumab 300 mg: Participants initially randomized to 300 mg risankizumab continued to receive 300 mg risankizumab SC at Week 16, Week 28, and Week 40 in Period B.
Period: Period A (Week 0 to Week 16)
Arm/Group | Period A: Placebo | Period A: Risankizumab 150 mg | Period A: Risankizumab 300 mg | Period B: Placebo / Risankizumab 150 mg | Period B: Placebo / Risankizumab 300 mg | Period B: Risankizumab 150 mg / Risankizumab 150 mg | Period B: Risankizumab 300 mg / Risankizumab 300 mg
Started (Randomized) | 34 | 69 | 69 | 0 | 0 | 0 | 0
Received Study Drug | 34 | 69 | 69 | 0 | 0 | 0 | 0
Completed (Competed Period A) | 25 | 61 | 58 | 0 | 0 | 0 | 0
Not Completed | 9 | 8 | 11 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 3 | 2 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrew Consent | 3 | 5 | 4 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 1 | 4 | 0 | 0 | 0 | 0
Not completed — Other | 2 | 0 | 2 | 0 | 0 | 0 | 0
Period: Period B (Week 16 to Week 52)
Arm/Group | Period A: Placebo | Period A: Risankizumab 150 mg | Period A: Risankizumab 300 mg | Period B: Placebo / Risankizumab 150 mg | Period B: Placebo / Risankizumab 300 mg | Period B: Risankizumab 150 mg / Risankizumab 150 mg | Period B: Risankizumab 300 mg / Risankizumab 300 mg
Started | 0 | 0 | 0 | 13 | 12 | 61 | 58
Received Study Drug | 0 | 0 | 0 | 13 | 11 | 61 | 57
Completed (Completed study) | 0 | 0 | 0 | 5 | 3 | 33 | 30
Not Completed | 0 | 0 | 0 | 8 | 9 | 28 | 28
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 2 | 3 | 0
Not completed — Withdrew Consent | 0 | 0 | 0 | 3 | 2 | 1 | 10
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 1 | 1
Not completed — Other | 0 | 0 | 0 | 4 | 5 | 23 | 17

BASELINE CHARACTERISTICS:
Population: The intent-to-treat population includes all randomized participants
Groups:
- Placebo: Participants randomized to receive placebo by subcutaneous (SC) injection at Weeks 0 and 4 in Period A.
- Risankizumab 150 mg: Participants randomized to receive 150 mg risankizumab SC at Weeks 0 and 4 in Period A.
- Risankizumab 300 mg: Participants randomized to receive 300 mg risankizumab SC at Weeks 0 and 4 in Period A.
- Total: Total of all reporting groups
Arm/Group | Placebo | Risankizumab 150 mg | Risankizumab 300 mg | Total
Number analyzed (Participants) | 34 | 69 | 69 | 172
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.5 (19.66) | 41.7 (15.12) | 43.8 (16.63) | 43.3 (16.66)
Age, Customized [Count of Participants; unit: Participants]
  < 18 years | 0 | 1 | 1 | 2
  18 - 39 years | 15 | 34 | 27 | 76
  40 - 64 years | 10 | 27 | 36 | 73
  ≥ 65 years | 9 | 7 | 5 | 21
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 31 | 32 | 76
  Male | 21 | 38 | 37 | 96
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 8 | 6 | 14
  Not Hispanic or Latino | 34 | 61 | 63 | 158
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 17 | 39 | 36 | 92
  Black or African American | 7 | 8 | 11 | 26
  Asian | 8 | 21 | 20 | 49
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1 | 2
  American Indian or Alaska Native | 0 | 1 | 1 | 2
  Multiple | 1 | 0 | 0 | 1
Geographic Region [Count of Participants; unit: Participants] — Rest of world includes United States, Puerto Rico, Canada, and Australia.
  Participants
    Japan | 6 | 13 | 13 | 32
    Rest of World | 28 | 56 | 56 | 140
Disease Severity [Count of Participants; unit: Participants] — Validated Investigator Global Assessment scale for Atopic Dermatitis (vIGA-AD) was used to assess the severity of AD based on lesion appearance on the following scale:
  * 0-Clear: No signs of AD;
  * 1-Almost clear: Barely perceptible erythema, induration/papulation and/or lichenification;
  * 2-Mild: Slight but definite erythema, induration/papulation and/or minimal lichenification. No oozing or crusting;
  * 3-Moderate: Clearly perceptible erythema, induration/papulation and/or lichenification, possible oozing or crusting;
  * 4-Severe: Marked erythema, induration/papulation and/or lichenification
  Participants
    3 (Moderate) | 20 | 40 | 39 | 99
    4 (Severe) | 14 | 29 | 30 | 73
Eczema Area and Severity Index (EASI) Score [Mean (Standard Deviation); unit: score on a scale] — EASI measures the extent and severity of atopic eczema based on assessments of the head/neck, trunk, upper limbs and lower limbs. For each region the percentage of skin affected and the severity (scored as none [0], mild [1], moderate [2], or severe [3]) for redness, thickness, scratching, and lichenification are assessed. The score for each region is calculated by multiplying the severity score by the area score, and adjusting for the proportion of the body region to the whole body. The EASI score is the sum of the scores for each region and ranges from 0 to 72 (worse disease).
  score on a scale | 30.85 (12.345) | 31.06 (13.995) | 28.70 (11.247) | 30.07 (12.605)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving At Least a 75% Reduction From Baseline in Eczema Area and Severity Index (EASI 75) at Week 16
Description: EASI is a tool used to measure the extent (area) and severity of atopic eczema based on assessments of the head/neck, trunk, upper limbs and lower limbs. For each region the area score is recorded as the percentage of skin affected by eczema. For each region, the severity score is calculated as the sum of the intensity scores (scored as none [0], mild [1], moderate [2], or severe [3]) for redness (erythema, inflammation), thickness (induration, papulation, swelling - acute eczema), scratching (excoriation), and lichenification (lined skin, prurigo nodules - chronic eczema).
  The total EASI score for each region is calculated by multiplying the severity score by the area score, with adjustment for the proportion of the body region to the whole body. The final EASI score is the sum of the 4 region scores and ranges from 0 to 72 where higher scores represent worse disease.
Time Frame: Baseline and Week 16
Population: Intent-to-treat population; non-responder imputation incorporating multiple imputation (MI) to handle missing data due to coronavirus pandemic 2019 (COVID-19) (NRI-C) was used in the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Risankizumab 150 mg | Risankizumab 300 mg
Number analyzed (Participants) | 34 | 69 | 69
percentage of participants | 11.8 [0.9 to 22.6] | 24.6 [14.5 to 34.8] | 21.7 [12.0 to 31.5]
Statistical Analysis 1: Comparison: Placebo vs Risankizumab 150 mg; Test type: Superiority; p = 0.084, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test stratified by Baseline disease severity (moderate [vIGA-AD 3] versus severe [vIGA-AD 4]); Adjusted Difference = 13.0, 95% CI 2-sided [-1.7 to 27.7] — Between Group Difference = Risankizumab - Placebo
Statistical Analysis 2: Comparison: Placebo vs Risankizumab 300 mg; Test type: Superiority; p = 0.179, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test stratified by Baseline disease severity (moderate [vIGA-AD 3] versus severe [vIGA-AD 4]); Adjusted Difference = 10.0, 95% CI 2-sided [-4.6 to 24.6] — Between Group Difference = Risankizumab - Placebo

2. Secondary Outcome: Percentage of Participants Who Achieved a vIGA-AD Score of "0" or "1" With a Reduction From Baseline of ≥ 2 Points at Week 16
Description: Validated Investigator Global Assessment scale for Atopic Dermatitis (vIGA-AD) was used to assess the severity of AD based on lesion appearance on the following scale:
  * 0 - Clear: No signs of AD;
  * 1 - Almost clear: Barely perceptible erythema, induration/papulation and/or lichenification;
  * 2 - Mild: Slight but definite erythema, induration/papulation and/or minimal lichenification. No oozing or crusting;
  * 3 - Moderate: Clearly perceptible erythema, induration/papulation and/or lichenification, possible oozing or crusting;
  * 4 - Severe: Marked erythema, induration/papulation and/or lichenification; possible oozing or crusting.
Time Frame: Baseline and Week 16
Population: Intent-to-treat population; non-responder imputation incorporating multiple imputation to handle missing data due to COVID-19 (NRI-C) was used in the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Risankizumab 150 mg | Risankizumab 300 mg
Number analyzed (Participants) | 34 | 69 | 69
percentage of participants | 5.9 [0.0 to 13.8] | 14.5 [6.2 to 22.8] | 5.8 [0.3 to 11.3]
Statistical Analysis 1: Comparison: Placebo vs Risankizumab 150 mg; Test type: Superiority; p = 0.129, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test stratified by Baseline disease severity (moderate [vIGA-AD 3] versus severe [vIGA-AD 4]); Adjusted Difference = 8.7, 95% CI 2-sided [-2.5 to 20.0] — Between Group Difference = Risankizumab - Placebo
Statistical Analysis 2: Comparison: Placebo vs Risankizumab 300 mg; Test type: Superiority; p = 0.994, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test stratified by Baseline disease severity (moderate [vIGA-AD 3] versus severe [vIGA-AD 4]); Adjusted Difference = -0.0, 95% CI 2-sided [-9.4 to 9.4] — Between Group Difference = Risankizumab - Placebo

3. Secondary Outcome: Percentage of Participants Who Achieved a Reduction of ≥ 4 Points in Worst Pruritus Numerical Rating Scale (NRS) Score From Baseline to Week 16
Description: Participants were asked to rate itch (pruritus) intensity at its worst during the past 24 hours on an 11-point scale from 0 (no itch) to 10 (worst imaginable itch).
Time Frame: Baseline and Week 16
Population: Intent-to-treat population with a Baseline Pruritus NRS of ≥ 4; non-responder imputation incorporating multiple imputation to handle missing data due to COVID-19 (NRI-C) was used in the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Risankizumab 150 mg | Risankizumab 300 mg
Number analyzed (Participants) | 33 | 66 | 66
percentage of participants | 0 [NA to NA] — Could not be calculated using the normal approximation to the binomial distribution | 13.6 [5.4 to 21.9] | 15.2 [6.5 to 23.8]
Statistical Analysis 1: Comparison: Placebo vs Risankizumab 150 mg; Test type: Superiority; p = 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test stratified by Baseline disease severity (moderate [vIGA-AD 3] versus severe [vIGA-AD 4]); Adjusted Difference = 13.7, 95% CI 2-sided [5.4 to 22.1] — Between Group Difference = Risankizumab - Placebo
Statistical Analysis 2: Comparison: Placebo vs Risankizumab 300 mg; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test stratified by Baseline disease severity (moderate [vIGA-AD 3] versus severe [vIGA-AD 4]); Adjusted Difference = 15.3, 95% CI 2-sided [6.6 to 24.0] — Between Group Difference = Risankizumab - Placebo

4. Secondary Outcome: Percent Change From Baseline in EASI Score at Week 16
Description: EASI is a tool used to measure the extent (area) and severity of atopic eczema based on assessments of the head/neck, trunk, upper limbs and lower limbs. For each region the area score is recorded as the percentage of skin affected by eczema. For each region, the severity score is calculated as the sum of the intensity scores (scored as none [0], mild [1], moderate [2], or severe [3]) for redness (erythema, inflammation), thickness (induration, papulation, swelling - acute eczema), scratching (excoriation), and lichenification (lined skin, prurigo nodules - chronic eczema).
  The total EASI score for each region is calculated by multiplying the severity score by the area score, with adjustment for the proportion of the body region to the whole body. The final EASI score is the sum of the 4 region scores and ranges from 0 to 72 where higher scores represent worse disease; a negative change from Baseline indicates improvement.
Time Frame: Baseline and Week 16
Population: Intent-to-treat population; missing data were handled using a mixed-effect model with repeated measurements (MMRM). The overall number of participants analyzed is based on the number of participants with non-missing Baseline and Week 16 values.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Risankizumab 150 mg | Risankizumab 300 mg
Number analyzed (Participants) | 17 | 51 | 43
percent change | -28.54 (9.378) | -38.86 (5.989) | -45.39 (6.351)
Statistical Analysis 1: Comparison: Placebo vs Risankizumab 150 mg; Test type: Superiority; p = 0.353, Mixed Effect Model Repeated Measurement; MMRM analysis with treatment, visit, treatment-by-visit interaction, vIGA-AD categories (moderate vs severe) and Baseline value in the model; Least Squares (LS) Mean Difference = -10.32, 95% CI 2-sided [-32.25 to 11.61], Standard Error of Mean 11.073 — Between Group Difference = Risankizumab - Placebo
Statistical Analysis 2: Comparison: Placebo vs Risankizumab 300 mg; Test type: Superiority; p = 0.139, Mixed Effect Model Repeated Measurement; [statistical method as in outcome 4, analysis 1]; LS Mean Difference = -16.86, 95% CI 2-sided [-39.24 to 5.53], Standard Error of Mean 11.305 — Between Group Difference = Risankizumab - Placebo

5. Secondary Outcome: Percent Change From Baseline in EASI Score at Week 28 and Week 52
Description: EASI is used to measure the extent (area) and severity of atopic eczema based on assessments of the head/neck, trunk, upper limbs and lower limbs. For each region the area score is recorded as the percentage of skin affected and the severity score is calculated as the sum of the intensity scores (scored as none [0], mild [1], moderate [2], or severe [3]) for redness (erythema, inflammation), thickness (induration, papulation, swelling), scratching, and lichenification (lined skin, prurigo nodules).
  The total EASI score for each region is calculated by multiplying the severity score by the area score, with adjustment for the proportion of the body region to the whole body. The final EASI score is the sum of the 4 region scores and ranges from 0 to 72 where higher scores represent worse disease; a negative change from Baseline indicates improvement.
  LS means were calculated from an analysis of covariance (ANCOVA) model with Baseline, treatment and vIGA-AD categories in the model.
Time Frame: Baseline and Weeks 28 and 52
Population: Intent-to-treat population with available data at each time point.
Measure: Least Squares Mean (Standard Error); unit: percent change
Groups:
- Placebo / Risankizumab 150 mg: Participants initially randomized to placebo were re-randomized at Week 16 to receive 150 mg risankizumab SC at Week 16, Week 28, and Week 40 in Period B.
- Placebo / Risankizumab 300 mg: Participants initially randomized to placebo were re-randomized at Week 16 to receive 300 mg risankizumab SC at Week 16, Week 28, and Week 40 in Period B.
- Risankizumab 150 mg / Risankizumab 150 mg: Participants initially randomized to 150 mg risankizumab in Period A continued to receive 150 mg risankizumab SC at Week 16, Week 28, and Week 40 in Period B.
- Risankizumab 300 mg / Risankizumab 300 mg: Participants initially randomized to 300 mg risankizumab in Period A continued to receive 300 mg risankizumab SC at Week 16, Week 28, and Week 40 in Period B.
Arm/Group | Placebo / Risankizumab 150 mg | Placebo / Risankizumab 300 mg | Risankizumab 150 mg / Risankizumab 150 mg | Risankizumab 300 mg / Risankizumab 300 mg
Number analyzed (Participants) | 8 | 5 | 45 | 43
percent change
  Week 28 | -58.60 (12.091) | -59.81 (14.956) | -62.44 (5.065) | -63.77 (5.051)
  Week 52: number analyzed (Participants) | 5 | 4 | 37 | 33
  Week 52 | -31.39 (12.979) | -76.75 (14.199) | -67.47 (4.663) | -62.70 (4.875)

6. Secondary Outcome: Percentage of Participants Who Achieved an EASI 75 Response at Week 28 and Week 52
Description: as for outcome 1
Time Frame: Baseline and Weeks 28 and 52
Population: Intent-to-treat population with available data at each time point.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo / Risankizumab 150 mg | Placebo / Risankizumab 300 mg | Risankizumab 150 mg / Risankizumab 150 mg | Risankizumab 300 mg / Risankizumab 300 mg
Number analyzed (Participants) | 8 | 5 | 45 | 43
percentage of participants
  Week 28 | 37.5 [4.0 to 71.0] | 0 [NA to NA] — Could not be calculated using the normal approximation to the binomial distribution | 53.3 [38.8 to 67.9] | 41.9 [27.1 to 56.6]
  Week 52: number analyzed (Participants) | 5 | 4 | 37 | 33
  Week 52 | 0 [NA to NA] — Could not be calculated using the normal approximation to the binomial distribution | 75.0 [32.6 to 100.0] | 43.2 [27.3 to 59.2] | 45.5 [28.5 to 62.4]

7. Secondary Outcome: Percentage of Participants Who Achieved an EASI 50 Response at Week 16
Description: EASI is a tool used to measure the extent (area) and severity of atopic eczema based on assessments of the head/neck, trunk, upper limbs and lower limbs. For each region the area score is recorded as the percentage of skin affected by eczema. For each region, the severity score is calculated as the sum of the intensity scores (scored as none [0], mild [1], moderate [2], or severe [3]) for redness (erythema, inflammation), thickness (induration, papulation, swelling - acute eczema), scratching (excoriation), and lichenification (lined skin, prurigo nodules - chronic eczema).
  The total EASI score for each region is calculated by multiplying the severity score by the area score, with adjustment for the proportion of the body region to the whole body. The final EASI score is the sum of the 4 region scores and ranges from 0 to 72 where higher scores represent worse disease.
  EASI 50 response is defined as at least a 50% reduction (improvement) from Baseline in EASI score.
Time Frame: Baseline and Week 16
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Risankizumab 150 mg | Risankizumab 300 mg
Number analyzed (Participants) | 34 | 69 | 69
percentage of participants | 29.4 [14.1 to 44.7] | 42.0 [30.4 to 53.7] | 34.8 [23.5 to 46.0]
Statistical Analysis 1: Comparison: Placebo vs Risankizumab 150 mg; Test type: Superiority; p = 0.171, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test stratified by Baseline disease severity (moderate [vIGA-AD 3] versus severe [vIGA-AD 4]); Adjusted Difference = 12.9, 95% CI 2-sided [-5.6 to 31.4] — Between Group Difference = Risankizumab - Placebo
Statistical Analysis 2: Comparison: Placebo vs Risankizumab 300 mg; Test type: Superiority; p = 0.552, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test stratified by Baseline disease severity (moderate [vIGA-AD 3] versus severe [vIGA-AD 4]); Adjusted Difference = 5.7, 95% CI 2-sided [-13.1 to 24.5] — Between Group Difference = Risankizumab - Placebo

8. Secondary Outcome: Percentage of Participants Who Achieved an EASI 50 Response at Week 28 and Week 52
Description: EASI is a tool used to measure the extent (area) and severity of atopic eczema based on assessments of the head/neck, trunk, upper limbs and lower limbs. For each region the area score is recorded as the percentage of skin affected by eczema. For each region, the severity score is calculated as the sum of the intensity scores (scored as none [0], mild [1], moderate [2], or severe [3]) for redness (erythema, inflammation), thickness (induration, papulation, swelling - acute eczema), scratching (excoriation), and lichenification (lined skin, prurigo nodules - chronic eczema).
  The total EASI score for each region is calculated by multiplying the severity score by the area score, with adjustment for the proportion of the body region to the whole body. The final EASI score is the sum of the 4 region scores and ranges from 0 to 72 where higher scores represent worse disease.
  An EASI 50 response is defined as at least a 50% reduction (improvement) from Baseline in EASI score.
Time Frame: Baseline and Weeks 28 and 52
Population: Intent-to-treat population with available data at each time point.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo / Risankizumab 150 mg | Placebo / Risankizumab 300 mg | Risankizumab 150 mg / Risankizumab 150 mg | Risankizumab 300 mg / Risankizumab 300 mg
Number analyzed (Participants) | 8 | 5 | 45 | 43
percentage of participants
  Week 28 | 75.0 [45.0 to 100.0] | 80.0 [44.9 to 100.0] | 73.3 [60.4 to 86.3] | 74.4 [61.4 to 87.5]
  Week 52: number analyzed (Participants) | 5 | 4 | 37 | 33
  Week 52 | 40.0 [0.0 to 82.9] | 75.0 [32.6 to 100.0] | 78.4 [65.1 to 91.6] | 72.7 [57.5 to 87.9]

9. Secondary Outcome: Percentage of Participants Who Achieved an EASI 90 Response at Week 16
Description: EASI is a tool used to measure the extent (area) and severity of atopic eczema based on assessments of the head/neck, trunk, upper limbs and lower limbs. For each region the area score is recorded as the percentage of skin affected by eczema. For each region, the severity score is calculated as the sum of the intensity scores (scored as none [0], mild [1], moderate [2], or severe [3]) for redness (erythema, inflammation), thickness (induration, papulation, swelling - acute eczema), scratching (excoriation), and lichenification (lined skin, prurigo nodules - chronic eczema).
  The total EASI score for each region is calculated by multiplying the severity score by the area score, with adjustment for the proportion of the body region to the whole body. The final EASI score is the sum of the 4 region scores and ranges from 0 to 72 where higher scores represent worse disease.
  An EASI 90 response is defined as at least a 90% reduction (improvement) from Baseline in EASI score.
Time Frame: Baseline, Week 16
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Risankizumab 150 mg | Risankizumab 300 mg
Number analyzed (Participants) | 34 | 69 | 69
percentage of participants | 2.9 [0.0 to 8.6] | 14.5 [6.2 to 22.8] | 8.7 [2.0 to 15.3]
Statistical Analysis 1: Comparison: Placebo vs Risankizumab 150 mg; Test type: Superiority; p = 0.022, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test stratified by Baseline disease severity (moderate [vIGA-AD 3] versus severe [vIGA-AD 4]); Adjusted Difference = 11.6, 95% CI 2-sided [1.7 to 21.6] — Between Group Difference = Risankizumab - Placebo
Statistical Analysis 2: Comparison: Placebo vs Risankizumab 300 mg; Test type: Superiority; p = 0.192, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test stratified by Baseline disease severity (moderate [vIGA-AD 3] versus severe [vIGA-AD 4]); Adjusted Difference = 5.8, 95% CI 2-sided [-2.9 to 14.4] — Between Group Difference = Risankizumab - Placebo

10. Secondary Outcome: Percentage of Participants Who Achieved an EASI 90 Response at Week 28 and Week 52
Description: as for outcome 9
Time Frame: Baseline and Weeks 28 and 52
Population: Intent-to-treat population with available data at each time point
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo / Risankizumab 150 mg | Placebo / Risankizumab 300 mg | Risankizumab 150 mg / Risankizumab 150 mg | Risankizumab 300 mg / Risankizumab 300 mg
Number analyzed (Participants) | 8 | 5 | 45 | 43
percentage of participants
  Week 28 | 25.0 [0.0 to 55.0] | 0 [NA to NA] — Could not be calculated using the normal approximation to the binomial distribution | 26.7 [13.7 to 39.6] | 27.9 [14.5 to 41.3]
  Week 52: number analyzed (Participants) | 5 | 4 | 37 | 33
  Week 52 | 0 [NA to NA] — Could not be calculated using the normal approximation to the binomial distribution | 0 [NA to NA] — Could not be calculated using the normal approximation to the binomial distribution | 24.3 [10.5 to 38.1] | 18.2 [5.0 to 31.3]

11. Secondary Outcome: Percentage of Participants Who Achieved a vIGA-AD Score of "0" or "1" With a Reduction From Baseline of ≥ 2 Points at Week 28 and Week 52
Description: as for outcome 2
Time Frame: Baseline and Weeks 28 and 52
Population: Intent-to-treat population with available data at each time point
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo / Risankizumab 150 mg | Placebo / Risankizumab 300 mg | Risankizumab 150 mg / Risankizumab 150 mg | Risankizumab 300 mg / Risankizumab 300 mg
Number analyzed (Participants) | 8 | 5 | 45 | 43
percentage of participants
  Week 28 | 0 [NA to NA] — Could not be calculated using the normal approximation to the binomial distribution | 0 [NA to NA] — Could not be calculated using the normal approximation to the binomial distribution | 22.2 [10.1 to 34.4] | 25.6 [12.5 to 38.6]
  Week 52: number analyzed (Participants) | 5 | 4 | 37 | 33
  Week 52 | 0 [NA to NA] — Could not be calculated using the normal approximation to the binomial distribution | 0 [NA to NA] — Could not be calculated using the normal approximation to the binomial distribution | 24.3 [10.5 to 38.1] | 21.2 [7.3 to 35.2]

12. Secondary Outcome: Change From Baseline in Percentage of Body Surface Area (BSA) Affected by Atopic Dermatitis at Week 16
Description: Body surface area (BSA) affected by atopic dermatitis was assessed by the physician and is expressed as a percentage of the total BSA. For purposes of the estimation, the total surface of the participant's palm plus five digits was assumed to be approximately equivalent to 1% BSA. A negative change from Baseline indicates improvement.
Time Frame: Baseline and Week 16
Population: Intent-to-treat population; missing data were handled using a mixed-effect model with repeated measurements. The overall number of participants analyzed is based on the number of participants with non-missing Baseline and Week 16 values.
Measure: Least Squares Mean (Standard Error); unit: percentage of body surface area
Arm/Group | Placebo | Risankizumab 150 mg | Risankizumab 300 mg
Number analyzed (Participants) | 17 | 51 | 43
percentage of body surface area | -7.41 (3.813) | -13.64 (2.429) | -13.27 (2.569)
Statistical Analysis 1: Comparison: Placebo vs Risankizumab 150 mg; Test type: Superiority; p = 0.169, Mixed Effect Model Repeated Measurement; [statistical method as in outcome 4, analysis 1]; LS Mean Difference = -6.24, 95% CI 2-sided [-15.15 to 2.68], Standard Error of Mean 4.506 — Between Group Difference = Risankizumab - Placebo
Statistical Analysis 2: Comparison: Placebo vs Risankizumab 300 mg; Test type: Superiority; p = 0.204, Mixed Effect Model Repeated Measurement; [statistical method as in outcome 4, analysis 1]; LS Mean Difference = -5.86, 95% CI 2-sided [-14.94 to 3.22], Standard Error of Mean 4.589 — Between Group Difference = Risankizumab - Placebo

13. Secondary Outcome: Change From Baseline in Percentage of BSA Affected by Atopic Dermatitis at Weeks 28 and 52
Description: Body surface area (BSA) affected by atopic dermatitis was assessed by the physician and is expressed as a percentage of the total BSA. For purposes of the estimation, the total surface of the participant's palm plus five digits was assumed to be approximately equivalent to 1% BSA. A negative change from Baseline indicates improvement.
  LS means and standard errors were calculated from ANCOVA with Baseline, treatment and stratum (Baseline vIGA-AD categories) in the model.
Time Frame: Baseline and Weeks 28 and 52
Population: Intent-to-treat population with available data at each time point
Measure: Least Squares Mean (Standard Error); unit: percentage of body surface area
Arm/Group | Placebo / Risankizumab 150 mg | Placebo / Risankizumab 300 mg | Risankizumab 150 mg / Risankizumab 150 mg | Risankizumab 300 mg / Risankizumab 300 mg
Number analyzed (Participants) | 8 | 5 | 45 | 43
percentage of body surface area
  Week 28 | -20.07 (5.843) | -11.90 (7.294) | -23.23 (2.438) | -23.22 (2.443)
  Week 52: number analyzed (Participants) | 5 | 4 | 37 | 33
  Week 52 | -0.86 (6.525) | -30.23 (7.316) | -29.26 (2.400) | -22.14 (2.510)

14. Secondary Outcome: Percentage of Participants Who Achieved a 50% Improvement in SCORing Atopic Dermatitis (SCORAD) Score (SCORAD 50) at Week 16
Description: SCORAD is a clinical tool used to assess the extent and severity of eczema (SCORing Atopic Dermatitis). The extent is assessed using the rule of 9 to calculate the affected area (A) as a percentage of the whole body (0-100%). The intensity part of the SCORAD (B) consists of 6 items: erythema, oedema/papulation, excoriations, lichenification, oozing/crusts and dryness, each graded on a scale from 0 (none) to 3 (severe), for a total score of 0 to 18. Subjective items (C) include daily pruritus and sleeplessness, each scored on a visual analogue scale (VAS) from 0 to 10 (total score 0-20). SCORAD is calculated as A/5 + 7B/2 + C, and ranges from 0 to 103 (worst).
Time Frame: Baseline, Week 16
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Risankizumab 150 mg | Risankizumab 300 mg
Number analyzed (Participants) | 34 | 69 | 69
percentage of participants | 18.0 [5.0 to 31.1] | 24.6 [14.5 to 34.8] | 13.0 [5.1 to 21.0]
Statistical Analysis 1: Comparison: Placebo vs Risankizumab 150 mg; Test type: Superiority; p = 0.422, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test stratified by Baseline disease severity (moderate [vIGA-AD 3] versus severe [vIGA-AD 4]); Adjusted Difference = 6.7, 95% CI 2-sided [-9.7 to 23.1] — Between Group Difference = Risankizumab - Placebo
Statistical Analysis 2: Comparison: Placebo vs Risankizumab 300 mg; Test type: Superiority; p = 0.505, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test stratified by Baseline disease severity (moderate [vIGA-AD 3] versus severe [vIGA-AD 4]); Adjusted Difference = -5.2, 95% CI 2-sided [-20.3 to 10.0] — Between Group Difference = Risankizumab - Placebo

15. Secondary Outcome: Percentage of Participants Who Achieved a SCORAD 50 Response at Week 28 and Week 52
Description: as for outcome 14
Time Frame: Baseline and Weeks 28 and 52
Population: Intent-to-treat population with available data at each time point.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo / Risankizumab 150 mg | Placebo / Risankizumab 300 mg | Risankizumab 150 mg / Risankizumab 150 mg | Risankizumab 300 mg / Risankizumab 300 mg
Number analyzed (Participants) | 9 | 5 | 46 | 43
percentage of participants
  Week 28 | 44.4 [12.0 to 76.9] | 20.0 [0.0 to 55.1] | 47.8 [33.4 to 62.3] | 37.2 [22.8 to 51.7]
  Week 52: number analyzed (Participants) | 6 | 4 | 38 | 37
  Week 52 | 0 [NA to NA] — Could not be calculated using the normal approximation to the binomial distribution | 50.0 [1.0 to 99.0] | 52.6 [36.8 to 68.5] | 35.1 [19.8 to 50.5]

16. Secondary Outcome: Percentage of Participants Who Achieved a SCORAD 75 Response at Week 16
Description: SCORAD is a clinical tool used to assess the extent and severity of eczema (SCORing Atopic Dermatitis). The extent is assessed using the rule of 9 to calculate the affected area (A) as a percentage of the whole body (0-100%). The intensity part of the SCORAD (B) consists of 6 items: erythema, oedema/papulation, excoriations, lichenification, oozing/crusts and dryness, each graded on a scale from 0 (none) to 3 (severe), for a total score of 0 to 18. Subjective items (C) include daily pruritus and sleeplessness, each scored on a visual analogue scale (VAS) from 0 to 10 (total score 0-20). SCORAD is calculated as A/5 + 7B/2 + C, and ranges from 0 to 103 (worst).
  A SCORAD 75 response is defined as at least a 75% reduction (improvement) from Baseline in SCORAD score.
Time Frame: Baseline and Week 16
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Risankizumab 150 mg | Risankizumab 300 mg
Number analyzed (Participants) | 34 | 69 | 69
percentage of participants | 0 [NA to NA] — Could not be calculated using the normal approximation to the binomial distribution | 10.1 [3.0 to 17.3] | 2.9 [0.0 to 6.9]
Statistical Analysis 1: Comparison: Placebo vs Risankizumab 150 mg; Test type: Superiority; p = 0.005, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test stratified by Baseline disease severity (moderate [vIGA-AD 3] versus severe [vIGA-AD 4]); Adjusted Difference = 10.1, 95% CI 2-sided [3.0 to 17.3] — Between Group Difference = Risankizumab - Placebo
Statistical Analysis 2: Comparison: Placebo vs Risankizumab 300 mg; Test type: Superiority; p = 0.151, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test stratified by Baseline disease severity (moderate [vIGA-AD 3] versus severe [vIGA-AD 4]); Adjusted Difference = 2.9, 95% CI 2-sided [-1.1 to 6.8] — Between Group Difference = Risankizumab - Placebo

17. Secondary Outcome: Percentage of Participants Who Achieved a SCORAD 75 Response at Week 28 and Week 52
Description: as for outcome 16
Time Frame: Baseline and Weeks 28 and 52
Population: Intent-to-treat population with available data at each time point.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo / Risankizumab 150 mg | Placebo / Risankizumab 300 mg | Risankizumab 150 mg / Risankizumab 150 mg | Risankizumab 300 mg / Risankizumab 300 mg
Number analyzed (Participants) | 9 | 5 | 46 | 43
percentage of participants
  Week 28 | 11.1 [0.0 to 31.6] | 0 [NA to NA] — Could not be calculated using the normal approximation to the binomial distribution | 23.9 [11.6 to 36.2] | 11.6 [2.0 to 21.2]
  Week 52: number analyzed (Participants) | 6 | 4 | 38 | 37
  Week 52 | 0 [NA to NA] — Could not be calculated using the normal approximation to the binomial distribution | 0 [NA to NA] — Could not be calculated using the normal approximation to the binomial distribution | 21.1 [8.1 to 34.0] | 13.5 [2.5 to 24.5]

18. Secondary Outcome: Percentage of Participants Who Achieved a SCORAD 90 Response at Week 16
Description: SCORAD is a clinical tool used to assess the extent and severity of eczema (SCORing Atopic Dermatitis). The extent is assessed using the rule of 9 to calculate the affected area (A) as a percentage of the whole body (0-100%). The intensity part of the SCORAD (B) consists of 6 items: erythema, oedema/papulation, excoriations, lichenification, oozing/crusts and dryness, each graded on a scale from 0 (none) to 3 (severe), for a total score of 0 to 18. Subjective items (C) include daily pruritus and sleeplessness, each scored on a visual analogue scale (VAS) from 0 to 10 (total score 0-20). SCORAD is calculated as A/5 + 7B/2 + C, and ranges from 0 to 103 (worst).
  A SCORAD 90 response is defined as at least a 90% reduction (improvement) from Baseline in SCORAD score.
Time Frame: Baseline and Week 16
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Risankizumab 150 mg | Risankizumab 300 mg
Number analyzed (Participants) | 34 | 69 | 69
percentage of participants | 0 [NA to NA] — Could not be calculated using the normal approximation to the binomial distribution | 5.8 [0.3 to 11.3] | 1.4 [0.0 to 4.3]
Statistical Analysis 1: Comparison: Placebo vs Risankizumab 150 mg; Test type: Superiority; p = 0.035, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test stratified by Baseline disease severity (moderate [vIGA-AD 3] versus severe [vIGA-AD 4]); Adjusted Difference = 5.9, 95% CI 2-sided [0.4 to 11.3] — Between Group Difference = Risankizumab - Placebo
Statistical Analysis 2: Comparison: Placebo vs Risankizumab 300 mg; Test type: Superiority; p = 0.311, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test stratified by Baseline disease severity (moderate [vIGA-AD 3] versus severe [vIGA-AD 4]); Adjusted Difference = 1.5, 95% CI 2-sided [-1.4 to 4.4] — Between Group Difference = Risankizumab - Placebo

19. Secondary Outcome: Percentage of Participants Who Achieved a SCORAD 90 Response at Week 28 and Week 52
Description: as for outcome 18
Time Frame: Baseline and Weeks 28 and 52
Population: Intent-to-treat population with available data at each time point.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo / Risankizumab 150 mg | Placebo / Risankizumab 300 mg | Risankizumab 150 mg / Risankizumab 150 mg | Risankizumab 300 mg / Risankizumab 300 mg
Number analyzed (Participants) | 9 | 5 | 46 | 43
percentage of participants
  Week 28 | 0 [NA to NA] — Could not be calculated using the normal approximation to the binomial distribution | 0 [NA to NA] — Could not be calculated using the normal approximation to the binomial distribution | 6.5 [0.0 to 13.7] | 4.7 [0.0 to 10.9]
  Week 52: number analyzed (Participants) | 6 | 4 | 38 | 37
  Week 52 | 0 [NA to NA] — Could not be calculated using the normal approximation to the binomial distribution | 0 [NA to NA] — Could not be calculated using the normal approximation to the binomial distribution | 15.8 [4.2 to 27.4] | 10.8 [0.8 to 20.8]

20. Secondary Outcome: Percentage of Participants Who Achieved a Dermatology Life Quality Index (DLQI) Score of "0" or "1" at Week 16
Description: The DLQI is a 10-item validated questionnaire used to assess the impact of AD disease symptoms and treatment on quality of life (QoL). It consists of 10 questions evaluating impact of skin diseases on different aspects of a participant's QoL over the prior week, including symptoms and feelings, daily activities, leisure, work or school, personal relationships, and the side effects of treatment. Each item is scored on a 4-point scale (0 = not at all/not relevant; 1 = a little; 2 = a lot; and 3 = very much).
  Item scores are added to provide a total score, ranging from 0 to 30, with higher scores indicating greater impairment of QoL. A score of 0 or 1 means that the disease has no effect at all.
Time Frame: Week 16
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Risankizumab 150 mg | Risankizumab 300 mg
Number analyzed (Participants) | 34 | 69 | 69
percentage of participants | 9.0 [0.0 to 18.8] | 8.7 [2.0 to 15.3] | 5.8 [0.3 to 11.3]
Statistical Analysis 1: Comparison: Placebo vs Risankizumab 150 mg; Test type: Superiority; p = 0.965, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test stratified by Baseline disease severity (moderate [vIGA-AD 3] versus severe [vIGA-AD 4]); Adjusted Difference = -0.3, 95% CI 2-sided [-12.0 to 11.5] — Between Group Difference = Risankizumab - Placebo
Statistical Analysis 2: Comparison: Placebo vs Risankizumab 300 mg; Test type: Superiority; p = 0.583, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test stratified by Baseline disease severity (moderate [vIGA-AD 3] versus severe [vIGA-AD 4]); Adjusted Difference = -3.1, 95% CI 2-sided [-14.3 to 8.1] — Between Group Difference = Risankizumab - Placebo

21. Secondary Outcome: Percentage of Participants Who Achieved a DLQI Score of "0" or "1" at Week 28 and Week 52
Description: as for outcome 20
Time Frame: Weeks 28 and 52
Population: Intent-to-treat population with available data at each time point
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo / Risankizumab 150 mg | Placebo / Risankizumab 300 mg | Risankizumab 150 mg / Risankizumab 150 mg | Risankizumab 300 mg / Risankizumab 300 mg
Number analyzed (Participants) | 9 | 5 | 49 | 44
percentage of participants
  Week 28 | 22.2 [0.0 to 49.4] | 20.0 [0.0 to 55.1] | 16.3 [6.0 to 26.7] | 13.6 [3.5 to 23.8]
  Week 52: number analyzed (Participants) | 5 | 4 | 36 | 32
  Week 52 | 20.0 [0.0 to 55.1] | 25.0 [0.0 to 67.4] | 13.9 [2.6 to 25.2] | 15.6 [3.0 to 28.2]

22. Secondary Outcome: Percentage of Participants Who Achieved a Children's Dermatology Life Quality Index (CDLQI) Score of "0" or "1" at Week 16
Description: The CDLQI is a 10-item, validated questionnaire used to assess the impact of AD disease symptoms and treatment on QoL. The CDLQI has been validated for use in individuals 4-16 years old. It consists of 10 questions assessing impact of skin diseases on different aspects of a patient's QoL over the prior week. The CDLQI items include symptoms and feelings, daily activities, leisure, school, relationships, sleep, and treatment. Each item is scored on a 4-point scale (0 = not at all; 1 = only a little; 2 = quite a lot; and 3 = very much). Item scores (0 to 3) are added to provide a total score range of 0 to 30; higher scores indicate greater impairment of QoL. A score of 0 or 1 means that the disease has no effect at all.
  In this study, the CDLQI was administered to participants who were < 16 years old at Baseline.
Time Frame: Week 16
Population: Intent-to-treat population < 16 years old at the Baseline visit; Non-responder imputation incorporating multiple imputation to handle missing data due to COVID-19 (NRI-C) was used in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Risankizumab 150 mg | Risankizumab 300 mg
Number analyzed (Participants) | 0 | 1 | 1
percentage of participants |  | 0 | 0

23. Secondary Outcome: Percentage of Participants Who Achieved a CDLQI Score of "0" or "1" at Week 28 and Week 52
Description: as for outcome 22
Time Frame: Weeks 28 and 52
Population: Intent-to-treat population < 16 years old at the Baseline visit with available data at each time point
Measure: Number; unit: percentage of participants
Arm/Group | Placebo / Risankizumab 150 mg | Placebo / Risankizumab 300 mg | Risankizumab 150 mg / Risankizumab 150 mg | Risankizumab 300 mg / Risankizumab 300 mg
Number analyzed (Participants) | 0 | 0 | 1 | 0
percentage of participants
  Week 28 |  |  | 0 |
  Week 52: number analyzed (Participants) | 0 | 0 | 0 | 0

24. Secondary Outcome: Percentage of Participants Who Achieved a Reduction in DLQI of ≥ 4 Points From Baseline at Week 16 Among Those With a DLQI ≥ 4 at Baseline
Description: The DLQI is a 10-item validated questionnaire used to assess the impact of AD disease symptoms and treatment on quality of life (QoL). It consists of 10 questions evaluating impact of skin diseases on different aspects of a participant's QoL over the prior week, including symptoms and feelings, daily activities, leisure, work or school, personal relationships, and the side effects of treatment. Each item is scored on a 4-point scale (0 = not at all/not relevant; 1 = a little; 2 = a lot; and 3 = very much).
  Item scores are added to provide a total score, ranging from 0 to 30, with higher scores indicating greater impairment of QoL.
  A change in DLQI score of at least 4 points is considered the minimum clinically important difference (MCID).
Time Frame: Baseline and Week 16
Population: Intent-to-treat population with a Baseline DLQI of ≥ 4; Non-responder imputation incorporating multiple imputation to handle missing data due to COVID-19 (NRI-C) was used in the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Risankizumab 150 mg | Risankizumab 300 mg
Number analyzed (Participants) | 32 | 64 | 64
percentage of participants | 25.6 [10.3 to 41.0] | 31.3 [19.9 to 42.6] | 37.5 [25.6 to 49.4]
Statistical Analysis 1: Comparison: Placebo vs Risankizumab 150 mg; Test type: Superiority; p = 0.539, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test stratified by Baseline disease severity (moderate [vIGA-AD 3] versus severe [vIGA-AD 4]); Adjusted Difference = 5.9, 95% CI 2-sided [-13.0 to 24.9] — Between Group Difference = Risankizumab - Placebo
Statistical Analysis 2: Comparison: Placebo vs Risankizumab 300 mg; Test type: Superiority; p = 0.213, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test stratified by Baseline disease severity (moderate [vIGA-AD 3] versus severe [vIGA-AD 4]); Adjusted Difference = 12.2, 95% CI 2-sided [-7.0 to 31.5] — Between Group Difference = Risankizumab - Placebo

25. Secondary Outcome: Percentage of Participants Who Achieved a Reduction in DLQI of ≥ 4 Points From Baseline at Week 28 and Week 52 Among Those With a DLQI ≥ 4 at Baseline
Description: as for outcome 24
Time Frame: Baseline and Weeks 28 and 52
Population: Intent-to-treat population with a Baseline DLQI of ≥ 4 and with available data at each time point.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo / Risankizumab 150 mg | Placebo / Risankizumab 300 mg | Risankizumab 150 mg / Risankizumab 150 mg | Risankizumab 300 mg / Risankizumab 300 mg
Number analyzed (Participants) | 9 | 5 | 45 | 51
percentage of participants
  Week 28 | 77.8 [50.6 to 100.0] | 40.0 [0.0 to 82.9] | 66.7 [52.9 to 80.4] | 68.3 [54.0 to 82.5]
  Week 52: number analyzed (Participants) | 5 | 4 | 33 | 30
  Week 52 | 60.0 [17.1 to 100.0] | 50.0 [1.0 to 99.0] | 63.6 [47.2 to 80.0] | 66.7 [49.8 to 83.5]

26. Secondary Outcome: Change From Baseline in DLQI Score at Week 16
Description: The DLQI is a 10-item validated questionnaire used to assess the impact of AD disease symptoms and treatment on quality of life (QoL). It consists of 10 questions evaluating impact of skin diseases on different aspects of a participant's QoL over the prior week, including symptoms and feelings, daily activities, leisure, work or school, personal relationships, and the side effects of treatment. Each item is scored on a 4-point scale (0 = not at all/not relevant; 1 = a little; 2 = a lot; and 3 = very much).
  Item scores are added to provide a total score, ranging from 0 to 30, with higher scores indicating greater impairment of QoL. A negative change from Baseline indicates improvement.
Time Frame: Baseline and Week 16
Population: as for outcome 12
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Risankizumab 150 mg | Risankizumab 300 mg
Number analyzed (Participants) | 17 | 49 | 41
score on a scale | -3.4 (1.55) | -3.4 (0.95) | -4.4 (1.03)
Statistical Analysis 1: Comparison: Placebo vs Risankizumab 150 mg; Test type: Superiority; p = 0.988, Mixed Effect Model Repeated Measurement; [statistical method as in outcome 4, analysis 1]; LS Mean Difference = 0.0, 95% CI 2-sided [-3.6 to 3.6], Standard Error of Mean 1.82 — Between Group Difference = Risankizumab - Placebo
Statistical Analysis 2: Comparison: Placebo vs Risankizumab 300 mg; Test type: Superiority; p = 0.594, Mixed Effect Model Repeated Measurement; [statistical method as in outcome 4, analysis 1]; LS Mean Difference = -1.0, 95% CI 2-sided [-4.7 to 2.7], Standard Error of Mean 1.86 — Between Group Difference = Risankizumab - Placebo

27. Secondary Outcome: Change From Baseline in DLQI Score at Week 28 and Week 52
Description: The DLQI is a 10-item validated questionnaire used to assess the impact of AD disease symptoms and treatment on quality of life (QoL). It consists of 10 questions evaluating impact of skin diseases on different aspects of a participant's QoL over the prior week, including symptoms and feelings, daily activities, leisure, work or school, personal relationships, and the side effects of treatment. Each item is scored on a 4-point scale (0 = not at all/not relevant; 1 = a little; 2 = a lot; and 3 = very much).
  Item scores are added to provide a total score, ranging from 0 to 30, with higher scores indicating greater impairment of QoL. A negative change from Baseline indicates improvement.
  LS means and standard errors were calculated from an ANCOVA model with Baseline, treatment and stratum (Baseline vIGA-AD categories) in the model.
Time Frame: Baseline and Weeks 28 and 52
Population: Intent-to-treat population with available data at each time point.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo / Risankizumab 150 mg | Placebo / Risankizumab 300 mg | Risankizumab 150 mg / Risankizumab 150 mg | Risankizumab 300 mg / Risankizumab 300 mg
Number analyzed (Participants) | 9 | 5 | 48 | 43
score on a scale
  Week 28 | -8.0 (2.06) | -5.3 (2.69) | -7.1 (0.87) | -7.3 (0.93)
  Week 52: number analyzed (Participants) | 5 | 4 | 36 | 32
  Week 52 | -4.5 (2.99) | -5.0 (3.30) | -7.7 (1.11) | -6.5 (1.18)

28. Secondary Outcome: Change From Baseline in CDLQI Score at Week 16
Description: The CDLQI is a 10-item, validated questionnaire used to assess the impact of AD disease symptoms and treatment on QoL. The CDLQI has been validated for use in individuals 4-16 years old. It consists of 10 questions assessing impact of skin diseases on different aspects of a patient's QoL over the prior week. The CDLQI items include symptoms and feelings, daily activities, leisure, school, relationships, sleep, and treatment. Each item is scored on a 4-point scale (0 = not at all; 1 = only a little; 2 = quite a lot; and 3 = very much). Item scores (0 to 3) are added to provide a total score range of 0 to 30; higher scores indicate greater impairment of QoL. A negative change from Baseline indicates improvement.
  In this study, the CDLQI was administered to participants who were < 16 years old at the Baseline visit.
Time Frame: Baseline and Week 16
Population: Intent-to-treat population < 16 years old at the Baseline visit; missing data were handled using a mixed-effect model with repeated measurements. The overall number of participants analyzed is based on the number of participants with non-missing Baseline and Week 16 values.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Risankizumab 150 mg | Risankizumab 300 mg
Number analyzed (Participants) | 0 | 1 | 0
score on a scale |  | -2.0 (NA) — Not calculated for N=1 |

29. Secondary Outcome: Change From Baseline in CDLQI Score at Week 28 and Week 52
Description: The CDLQI is a 10-item, validated questionnaire used to assess the impact of AD disease symptoms and treatment on QoL. The CDLQI has been validated for use in individuals 4-16 years old. It consists of 10 questions assessing impact of skin diseases on different aspects of a patient's QoL over the prior week. The CDLQI items include symptoms and feelings, daily activities, leisure, school, relationships, sleep, and treatment. Each item is scored on a 4-point scale (0 = not at all; 1 = only a little; 2 = quite a lot; and 3 = very much). Item scores (0 to 3) are added to provide a total score range of 0 to 30; higher scores indicate greater impairment of QoL. A negative change from Baseline indicates improvement.
  In this study, the CDLQI was administered to participants who were < 16 years old at the Baseline visit.
  LS means were calculated from ANCOVA with Baseline and treatment in the model.
Time Frame: Baseline and Weeks 28 and 52
Population: Intent-to-treat population < 16 years old at the Baseline visit with available data at each time point.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo / Risankizumab 150 mg | Placebo / Risankizumab 300 mg | Risankizumab 150 mg / Risankizumab 150 mg | Risankizumab 300 mg / Risankizumab 300 mg
Number analyzed (Participants) | 0 | 0 | 1 | 0
score on a scale
  Week 28 |  |  | 1.0 (0.00) |
  Week 52: number analyzed (Participants) | 0 | 0 | 0 | 0

30. Secondary Outcome: Change From Baseline in Worst Pruritus Numerical Rating Scale at Week 16
Description: Participants were asked to rate itch (pruritus) intensity at its worst during the past 24 hours on an 11-point scale from 0 (no itch) to 10 (worst imaginable itch). Change from Baseline was calculated from a rolling weekly average. A negative change from Baseline indicates improvement.
Time Frame: Baseline and Week 16
Population: as for outcome 12
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Risankizumab 150 mg | Risankizumab 300 mg
Number analyzed (Participants) | 17 | 45 | 39
score on a scale | -0.098 (0.5110) | -1.416 (0.3408) | -1.746 (0.3619)
Statistical Analysis 1: Comparison: Placebo vs Risankizumab 150 mg; Test type: Superiority; p = 0.033, Mixed Effect Model Repeated Measurement; [statistical method as in outcome 4, analysis 1]; LS Mean Difference = -1.318, 95% CI 2-sided [-2.531 to -0.105], Standard Error of Mean 0.6137 — Between Group Difference = Risankizumab - Placebo
Statistical Analysis 2: Comparison: Placebo vs Risankizumab 300 mg; Test type: Superiority; p = 0.009, Mixed Effect Model Repeated Measurement; [statistical method as in outcome 4, analysis 1]; LS Mean Difference = -1.648, 95% CI 2-sided [-2.885 to -0.411], Standard Error of Mean 0.6260 — Between Group Difference = Risankizumab - Placebo

31. Secondary Outcome: Change From Baseline in Worst Pruritus NRS Score at Week 28 and Week 52
Description: Participants were asked to rate itch (pruritus) intensity at its worst during the past 24 hours on an 11-point scale from 0 (no itch) to 10 (worst imaginable itch). Change from Baseline was calculated from a rolling weekly average. A negative change from Baseline indicates improvement.
  LS means and standard errors were calculated from an ANCOVA with Baseline, treatment and stratum (Baseline vIGA-AD categories) in the model.
Time Frame: Baseline and Weeks 28 and 52
Population: Intent-to-treat population with available data at each time point.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo / Risankizumab 150 mg | Placebo / Risankizumab 300 mg | Risankizumab 150 mg / Risankizumab 150 mg | Risankizumab 300 mg / Risankizumab 300 mg
Number analyzed (Participants) | 9 | 5 | 50 | 44
score on a scale
  Week 28 | -2.685 (0.9303) | -3.182 (1.2347) | -2.474 (0.3887) | -2.684 (0.4179)
  Week 52: number analyzed (Participants) | 5 | 4 | 36 | 32
  Week 52 | -2.668 (1.2153) | -4.012 (1.3907) | -2.936 (0.4567) | -2.454 (0.4957)

32. Secondary Outcome: Percentage of Participants Who Achieved a Reduction of ≥ 4 Points From Baseline in Worst Pruritus NRS Score at Week 28 and Week 52
Description: as for outcome 3
Time Frame: Baseline and Weeks 28 and 52
Population: Intent-to-treat population with a Baseline Pruritus NRS of ≥ 4, and with available data at each time point.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo / Risankizumab 150 mg | Placebo / Risankizumab 300 mg | Risankizumab 150 mg / Risankizumab 150 mg | Risankizumab 300 mg / Risankizumab 300 mg
Number analyzed (Participants) | 9 | 5 | 48 | 43
percentage of participants
  Week 28 | 22.2 [0.0 to 49.4] | 20.0 [0.0 to 55.1] | 31.3 [18.1 to 44.4] | 39.5 [24.9 to 54.1]
  Week 52: number analyzed (Participants) | 5 | 4 | 34 | 32
  Week 52 | 20.0 [0.0 to 55.1] | 25.0 [0.0 to 67.4] | 38.2 [21.9 to 54.6] | 28.1 [12.5 to 43.7]

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to 20 weeks after last dose. Period A: 16 weeks for participants who entered Period B or up to 36 weeks for participants who did not enter Period B. Period B: From Week 16 up to Week 60.
Groups:
- Period A: Placebo: Participants received placebo by subcutaneous injection at Week 0 and Week 4 in Period A.
- Period A: Risankizumab 150 mg: Participants received 150 mg risankizumab SC at Week 0 and Week 4 in Period A.
- Period A: Risankizumab 300 mg: Participants received 300 mg risankizumab SC at Week 0 and Week 4 in Period A.
- Period B: Placebo / Risankizumab 150 mg: Participants initially randomized to placebo received 150 mg risankizumab SC at Week 16, Week 28, and Week 40 in Period B.
- Period B: Placebo / Risankizumab 300 mg: Participants initially randomized to placebo received 300 mg risankizumab SC at Week 16, Week 28, and Week 40 in Period B.
- Period B: Risankizumab 150 mg / Risankizumab 150 mg: Participants initially randomized to 150 mg risankizumab in Period A received 150 mg risankizumab SC at Week 16, Week 28, and Week 40 in Period B.
- Period B: Risankizumab 300 mg / Risankizumab 300 mg: Participants initially randomized to 300 mg risankizumab in Period A received 300 mg risankizumab SC at Week 16, Week 28, and Week 40 in Period B.
Arm/Group | Period A: Placebo | Period A: Risankizumab 150 mg | Period A: Risankizumab 300 mg | Period B: Placebo / Risankizumab 150 mg | Period B: Placebo / Risankizumab 300 mg | Period B: Risankizumab 150 mg / Risankizumab 150 mg | Period B: Risankizumab 300 mg / Risankizumab 300 mg
All-Cause Mortality (participants affected / at risk) | 1/34 | 0/69 | 0/69 | 0/13 | 0/11 | 0/61 | 0/57
Serious Adverse Events (participants affected / at risk) | 3/34 | 0/69 | 0/69 | 0/13 | 0/11 | 2/61 | 3/57
Other Adverse Events (participants affected / at risk) | 17/34 | 25/69 | 25/69 | 6/13 | 5/11 | 13/61 | 10/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Period A: Placebo (N=34) | Period A: Risankizumab 150 mg (N=69) | Period A: Risankizumab 300 mg (N=69) | Period B: Placebo / Risankizumab 150 mg (N=13) | Period B: Placebo / Risankizumab 300 mg (N=11) | Period B: Risankizumab 150 mg / Risankizumab 150 mg (N=61) | Period B: Risankizumab 300 mg / Risankizumab 300 mg (N=57)
ARRHYTHMIA (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
AMAUROSIS FUGAX (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CELLULITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
FRACTURED COCCYX (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SPINAL FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CERVIX CARCINOMA STAGE I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DERMATITIS ATOPIC (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Period A: Placebo (N=34) | Period A: Risankizumab 150 mg (N=69) | Period A: Risankizumab 300 mg (N=69) | Period B: Placebo / Risankizumab 150 mg (N=13) | Period B: Placebo / Risankizumab 300 mg (N=11) | Period B: Risankizumab 150 mg / Risankizumab 150 mg (N=61) | Period B: Risankizumab 300 mg / Risankizumab 300 mg (N=57)
LEUKOPENIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
BUNDLE BRANCH BLOCK RIGHT (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DENTAL CARIES (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
TOOTHACHE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
OEDEMA PERIPHERAL (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NASOPHARYNGITIS (Infections and infestations) | 0 (0) | 4 (6) | 4 (4) | 0 (0) | 0 (0) | 4 (4) | 3 (4)
SKIN INFECTION (Infections and infestations) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
TONSILLITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
TOOTH INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 2 (2) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
VIRAL UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BLOOD GLUCOSE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
BLOOD THYROID STIMULATING HORMONE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DIZZINESS POSTURAL (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
AMENORRHOEA (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ACNE (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DERMATITIS ATOPIC (Skin and subcutaneous tissue disorders) | 7 (7) | 19 (19) | 16 (16) | 2 (2) | 1 (1) | 7 (7) | 5 (5)
HYPERTROPHIC SCAR (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PRURITUS (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 5 (5) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
URTICARIA (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
WISDOM TEETH REMOVAL (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HYPERTENSION (Vascular disorders) | 3 (3) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2020-10-13): https://cdn.clinicaltrials.gov/large-docs/40/NCT03706040/Prot_000.pdf
  • Statistical Analysis Plan (2020-10-14): https://cdn.clinicaltrials.gov/large-docs/40/NCT03706040/SAP_001.pdf